CLINICAL TRIAL: NCT06512909
Title: Examining the Effects of Virtual Reality Glasses and Stress Ball Application on Pain, Anxiety and Patient Satisfaction in Intramuscular Injection Application: Randomized Controlled Study
Brief Title: Effects of Virtual Reality Glasses and Stress Ball Application on Pain, Anxiety and Patient Satisfaction in Intramuscular Injection Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Asude GÜNEY, Research Asisstant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Necmettin Üniversitesi
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pain and Anxiety During Intramuscular Injection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Voluntary Information and Consent Form, Patient Information Form and Visual Analogue Anxiety Scale will be filled out.
  Standard injection practice will be applied. Visual Comparison Scale (VAS-VAS), Satisfaction Assessment Scale (MDS) and Visual Analog Anxiety Scale (VAS-A) will be filled out within one minute after the procedure.
- Virtual Reality Glasses (Experimental): Voluntary Information and Consent Form, Patient Information Form and Visual Analogue Anxiety Scale will be filled out.
  The individual will be shown a video containing relaxing nature images via VR. Intramuscular injection will begin three minutes after the individual starts watching the video, and the procedure will be performed while continuing to watch the video. Visual Comparison Scale (VAS-VAS), Satisfaction Assessment Scale (MDS) and Visual Analog Anxiety Scale (VAS-A) will be completed within one minute after the procedure.
  Interventions: Other: Virtual Reality Glasses Application
- Stress ball (Experimental): Voluntary Information and Consent Form, Patient Information Form and Visual Analogue Anxiety Scale will be filled out.
  The individual will be given a stress ball on the side where the intramuscular injection will be administered. Three minutes after the individual starts squeezing the ball, the intramuscular injection will begin and the procedure will be performed while squeezing the ball. Visual Comparison Scale (VAS-VAS), Satisfaction Assessment Scale (MDS) and Visual Analog Anxiety Scale (VAS-A) will be filled out within one minute after the procedure.
  Interventions: Other: Stress Ball Application

INTERVENTIONS:
Other: Virtual Reality Glasses Application — A video containing relaxing nature images will be shown to a group via VR. Intramuscular injection will begin three minutes after the individual starts watching the video, and the procedure will be performed while continuing to watch the video.
  Arms: Virtual Reality Glasses
Other: Stress Ball Application — One group will be given a stress ball in the hand on the side where the intramuscular injection will be administered. Three minutes after the individual starts squeezing the ball, intramuscular injection will begin and the procedure will be performed while squeezing the ball.
  Arms: Stress ball

SUMMARY:
Purpose: This study was planned to examine the effects of virtual reality glasses and stress ball application on pain, anxiety and patient satisfaction in intramuscular injection application.

Material method: The data of the research were collected using "Sociodemographic Characteristics Form", "Visual Comparison Scale (VAS-VAS)", "Satisfaction Assessment Scale (MDS)" and "Visual Analog Anxiety Scale (VAS-A)". will be collected using .

Results: Findings will be presented in tables. Conclusion and recommendations: As a result, it is expected that the use of stress balls and virtual reality glasses in intramuscular application will be positive.

DETAILED DESCRIPTION:
Medication management is one of the basic nursing functions and these practices require knowledge and skills. Nurses administer medications via enteral and parenteral routes within the scope of their therapeutic roles. Among these applications, intravenous, subcutaneous, intradermal and intramuscular (IM) drug applications are parenteral drug application methods and are among the application authority of nurses. IM injection is defined as administering the drug deep into muscle tissue. IM injection can be applied from four different regions: deltoid, ventrogluteal, laterofemoral and femoral. The nurse will decide which area will be injected; It decides by taking into account the patient's body mass index, amount of medication, muscle development and muscle ratio. In injection applications, trauma caused by the needle while entering the tissue, not keeping the angle of entry into the tissue constant, the patient's previous experiences and psychological factors related to the patient may cause pain and affect the patient-nurse relationship, patient care quality and patient satisfaction.Nurses can reduce the individual's injection-related pain with the correct injection technique. In the literature, it is stated that nurses use local anesthetic creams and oral tablets pharmacologically during invasive procedures, while non-pharmacologically they use music therapy, vibrating tourniquet, buzzy device, various palpation techniques (Helfer Skin Tap Technique, etc.), therapeutic touch, stress ball and It has been stated that they use various distraction techniques such as virtual reality glasses. It is seen that the frequency of use of virtual reality, one of these methods, has increased in recent years with the developments in the technological field.

Virtual reality causes something or a situation that does not actually exist to be felt as real by creating it in three dimensions with computers and other tools. It is if he or she is really present in the created world. Studies have found that virtual reality glasses are effective on pain and anxiety in different groups and in different invasive applications. One of the methods of diverting attention in pain and anxiety management is the application of a stress ball, which is one of the methods aimed at the sense of touch. Stress ball is an application based on the pain theory that focuses on cognitive pain and anxiety management and reduces attention to painful stimuli by drawing attention to a different area. In stress ball application, the perception of pain is reduced due to the increased mental orientation towards more salient stimuli, and therefore the level of anxiety decreases. The stress ball is a simple, reliable, inexpensive and easily accessible application that helps reduce patients' anxiety. The stress ball, which is one of the applications to divert attention, is also an effective method to ensure cognitive focus. In the literature, it is seen that stress ball application is generally used to reduce pain and anxiety. There is no study in the literature comparing virtual reality glasses and stress ball application in intramuscular injection application. This study was planned to examine the effects of virtual reality glasses and stress ball application on pain, anxiety and patient satisfaction in intramuscular injection application.

H.4.1. Research Questions/Hypotheses: H1a: Virtual reality glasses, stress balls and intramuscular injections applied with standard methods affect patients' pain sensation at different levels. H1b: Virtual reality glasses, stress balls and intramuscular injections applied with standard methods affect patients' anxiety at different levels. H1c: Virtual reality glasses, stress balls and intramuscular injections applied with standard methods affect patients' satisfaction at different levels. Research Type: This research was planned as a triple blind-randomized controlled study. Place and Time of the Research: The research will be conducted with patients who applied to Meram Medical Faculty Hospital Emergency Department for treatment in July-August 2024. 35 nurses, 6 specialist physicians and 21 assistant physicians work in the emergency department. The emergency room consists of triage, isolation, trauma room, resuscitation, yellow area, green area, red area and special rooms. There is a stretcher in the triage room. In addition to 30 stretchers, there are 11 emergency observation, 5 intermediate intensive care and 9 critical care unit beds in the emergency department. There are two stretchers in the green area. Population and Sample of the Study: The population of the study will consist of patients who applied to the trauma area of Meram Medical Faculty Hospital Emergency Service between July and August 2024 to receive intramuscular tetanus vaccination. Before determining the sample of the study, a priori power analysis was performed in the GPOWER 3.1.9.7 Package Program based on analysis of variance in repeated measurements. It was determined that the number of samples required to exceed 90% of the power of the study with a 95% confidence interval, a significance level of 0.05 and a medium effect size was 108. Considering the possibility of data loss for various reasons, it was planned to include 120 patients in the study sample who met the research criteria (40: Control, 40: Virtual reality, 40: Stress ball).

Randomization: The study group of the research will be determined according to the inclusion and exclusion criteria. Patients who agree to participate in the study will be divided into three groups: two intervention groups and a control group. Patients will be randomly assigned to three groups: intervention-virtual reality glasses group, intervention-ball squeezing group, and control group. The assignment of patients to groups will be determined by the clinic nurse by drawing lots. Preliminary tests of the research will be applied after obtaining written consent from patients who meet the research criteria and agree to participate in the research. After the preliminary tests are administered, patients will be assigned to control and intervention groups by block randomization method.

Data Collection Tools Used in the Research The data of the research will be collected using the "Sociodemographic Characteristics Form", "Visual Comparison Scale (VAS-VAS)", Satisfaction Assessment Scale (MDS)" and "Visual Analog Anxiety Scale (VAS-A)".

Patient Information Form: This form was prepared using the researchers' experiences and literature. It consists of 9 questions such as age, gender, marital status, educational status, occupation, body mass index, experience of intramuscular injection into the deltoid muscle, presence of fear of injection, history of not giving injections or postponing injections. Visual Comparison Scale-Visual Analog Scale (VAS): The VAS scale is a unidimensional scale widely used today to assess pain intensity. Validity and reliability studies have been conducted for Türkiye. According to VAS, pain intensity was rated as 0 points as "no pain" and 10 points as "worst pain imaginable". Pain intensity ranges determined by VAS; A score below 3 points was determined as mild pain, between 3 and 6 points as moderate pain, and above 6 points as severe pain. The VAS scale will be administered to patients within 1 minute after injection to determine the severity of pain they feel during intramuscular injection. Satisfaction Rating Scale (MDS): Satisfaction of the patients after the injection was evaluated using a scale consisting of a 100 mm long vertical line with the words "Very Satisfied" at one end and "Very Dissatisfied" at the other end. Patients' satisfaction will be evaluated within 1 minute after the injection.

Visual Analog Anxiety Scale (VAS-A): It is a measurement tool that is 10 cm long, represents "no anxiety" as 0 points, "I feel a lot of anxiety" as 10 points, and is scored between 0-10. As the patient's anxiety level approaches 10, it indicates that his anxiety increases. It has been reported in the literature that it is a successful scale in relieving patients' symptoms and evaluating fast-acting drug treatments. There is a concurrent validity correlation between the VAS-A and the Spielberger State Anxiety Inventory (r=0.4916 to r=0.8219). This shows that although the VAS-A scale is short, it is a reliable and accurate measurement tool. The VAS-A scale will be administered to patients before and immediately after the injection. Data Collection: Data will be collected from patients admitted to the trauma area at the emergency department of Necmettin Erbakan University Faculty of Medicine Hospital. While data is being collected; The patient will be interviewed, informed about the research, and written consent will be obtained from the patient. Each patient will receive a tetanus shot only once. A nurse will work with the researcher during the procedure. All injections will be administered by the same nurse. Virtual reality glasses and stress ball interventions will be applied in the research.

Application tools: Virtual Reality Glasses (VR): VR glasses help people get away from the environment they are in and focus their attention on the image or sound by watching the content and/or listening with headphones. Thanks to the special lenses inside the glasses, the image is shown large and clear. With the Bluetooth stereo headset feature of the glasses, it is possible to block out ambient sounds and listen to the contents watched by the individual. Thus, the person experiences the feeling of being in a different environment by drawing his attention in a different direction thanks to the virtual environment he watches with virtual glasses. When watching content loaded on a smartphone with virtual reality glasses, the glasses easily provide the viewfinder distance required for panoramic vision by dividing the image into two equal windows. Head-mounted VR glasses can be personalized thanks to their adjustable straps. In particular, the distance between the mobile phone and the lens is fixed according to the individual. VR glasses have air vents that can dissipate the heat emitted by the smartphone. When using glasses, there is no need for any power or connection unit other than the phone. The smartphone's internet connection is only required to watch the content. An Oculus Quest-2 VR headset will be used in the research. These VR glasses are compatible with smartphones (Android, IOS). To use the glasses, the Meta Quest program will be downloaded to researchers' mobile phones. VR content will be selected from 3600 angle footage from YouTube.

Stress Ball: A stress ball is a soft toy, usually no larger than 7 cm, that is stuck in the hand and manipulated with the fingers to relieve stress and muscle tension, or to exercise the muscles. In addition to reducing stress, it is also used in physical therapy. Some stress balls are made from closed-cell polyurethane foam. Polyurethane is frequently preferred in the use of stress balls due to its ability to immediately return to its original shape. In this study, a stress ball with a flat surface, seven cm in diameter, made of soft material, can be squeezed in the hand, and returns to its original state when squeezed and released, will be used.

Research Variables Dependent variables: • Visual Comparison Scale mean score • Satisfaction Evaluation Scale mean score • Visual Analogue Anxiety Scale mean score Independent variables: • Sociodemographic Characteristics • Virtual reality and ball squeezing method Ethical Dimension of the Research: Subjects of the research, purpose, duration, plan, Where and how the data will be used will be explained to the patients included in the study. In line with the principles of volunteering and willingness, verbal and written consent will be obtained by reading the "Voluntary Information and Consent Form". In line with the principle of autonomy, patients and their relatives will be informed that they can withdraw from the study at any time, regardless of whether there is a reason to do so. Permission will be obtained from the institution where the research will be conducted and the nurse who will work in the clinic will be informed about the research. Limitations of the Study: The study is limited to patients who will be administered intramuscular tetanus vaccine by applying to the trauma area at the emergency department of Necmettin Erbakan University Faculty of Medicine Hospital. The data obtained as a result of the research can be generalized to this group. Statistical Evaluation of Data: Data will be analyzed with IBM SPSS 22 package program. For quantitative data, mean, standard deviation, median, interquartile range, minimum and maximum values, categorical data will be presented as frequency (percentage). The suitability of the data for normal distribution will be determined. Chi-square test, Kruskal Wallis test, Analysis of Variance and t test will be used in independent groups to compare categorical variables according to groups. It will be used in Tukey and Scheffe posthoc analyses. The significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Having a body mass index (BMI) between 18.5 and 30,
* No scar, incision, lipodystrophy or infection at the injection site
* Pain, fear etc. Not having any disease that prevents perception of variables (loss of vision, hearing, sensation, cognitive impairment, stroke, diabetes mellitus, etc.)
* Not using centrally or peripherally acting analgesics or sedatives,
* No deficiency in arm limbs,
* No sensory or motor deficits,
* No history of diabetes,
* No vision, hearing or perception problems,
* Being oriented to place and time,
* Volunteering to participate in the research.

Exclusion Criteria:

* Development of drug-related allergy or other complications
* Wants to withdraw from the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Visual Comparison Scale-Assessing pain with Visual Analog Scale | 1 minute after application
  According to VAS, pain intensity is rated as "no pain" as 0 points and "the worst pain imaginable" as 10 points (Eti Aslan, 2002). Pain intensity ranges determined by VAS; A score below 3 points was defined as mild pain, between 3 and 6 points as moderate pain, and above 6 points as severe pain.
Assessing anxiety level with the Visual Analog Anxiety Scale | Before application and 1 minute after application
  It is a measurement tool with a length of 10 cm, representing 0 points for "no anxiety" and 10 points for "I feel a lot of anxiety", and its evaluation is scored between 0-10. As the patient's anxiety level approaches 10, it indicates that his anxiety increases.
Evaluating patient satisfaction with the Satisfaction Rating Scale | 1 minute after application
  Patients' post-injection satisfaction was evaluated using a scale consisting of a 100 mm long vertical line with the words "Very Satisfied" on one end and "Not at all satisfied" on the other end.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)